CLINICAL TRIAL: NCT01168843
Title: Computer Program for Evaluation of the Symmetry Between the Primary Sulci of the Two Fetal Brain Hemispheres and Midsagittal Fetal Head Biometry Using 3-dimensional Ultrasound Planes.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Zvi Leibovitz, Bnai Zion medical center
Other Study IDs: 0027-10-BNZ
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-07

CONDITIONS: Normal Fetal Brain Sulcation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- normal pregnant
  Interventions: Other: computerized analysis of sonographic images

INTERVENTIONS:
Other: computerized analysis of sonographic images — Evaluation of the Symmetry between the Primary Sulci of the Two Fetal Brain Hemispheres Using 3-dimensional Ultrasound Planes

SUMMARY:
Computer Program for Evaluation of the Symmetry between the Primary Sulci of the Two Fetal Brain Hemispheres Using 3-dimensional Ultrasound Planes

This retrospective study is based on the computerized analysis of the orthogonal fetal brain planes.

The images are obtained from the digital archive of the fetal sonographic examinations done in Bnai Zion Medical Center.

In addition, midsagittal measurements of fetal head will be obtained from this archive of 3-dimensional images.

Study measurements will provide the quantitative parameters of normal fetal brain sulcation. Normal fetal head growth in midsagittal plane will be studied also.

ELIGIBILITY:
Inclusion Criteria:

* normal pregnancies
* proper dating

Exclusion Criteria:

* complications of pregnancy
* fetal malformations

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: normal pregnancies in 2nd and 3rd trimester
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-10

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel